CLINICAL TRIAL: NCT01143428
Title: Oxidative Stress in Motor Neuron Disease: COSMOS-PLS Add-On Study
Brief Title: Oxidative Stress in Motor Neuron Disease: COSMOS Add-On Study
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100121; 10-N-0121
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2019-11-05 (Actual); Status verified 2015-08-03

CONDITIONS: Motor Neuron Disease; Primary Lateral Sclerosis
Keywords: Motor Neuron Disease; Primary Lateral Sclerosis; Oxidative Stress; Physiology; PLS
MeSH Terms: conditions — Motor Neuron Disease

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

- Primary lateral sclerosis (PLS) is a disorder in which nerve cells in the brain that control movement degenerate. The cause of PLS is not known, but some research has suggested that environmental factors that produce oxidative stress trigger PLS in people who carry certain genes. Oxidative stress is caused when the body makes chemicals called "free radicals" faster than its natural systems can break them down. Oxidative stress can be triggered by exposures to chemicals related to the bodily effects of lead, smoking, alcohol consumption, physical activity, and psychological stress. Chemicals produced by the body during oxidative stress can be measured in the blood and urine. Researchers are interested in studying the physical, neurological, and chemical effects of PLS to better understand the effects of oxidative stress on the disorder.

Objectives:

- To study the relation of oxidative stress to the diagnosis and progression of motor neuron disease.

Eligibility:

- Individuals 20 years of age or older who have been diagnosed with PLS, and have had symptoms of PLS for at least 5 but not more than 8 years and been previously enrolled in 01-N-0145 Screening: Neurologic Disorders with Muscle Stiffness

Design:

* Participants will have an initial study visit and three follow-up visits. Each visit will require approximately 3 days of testing at the National Institutes of Health Clinical Center.
* As part of this study, participants will have the following tests and procedures:
* Neurological examination to test muscle strength, sensation, coordination, and reflexes, as well as clarity of speech
* Tests of memory, attention, concentration, and thinking
* Surveys on oxidative stress, including questions on life, mood, jobs held, and habit
* Electromyography to record the electrical activity of muscles
* Transcranial magnetic stimulation to measure electrical activity translated from their brain to the muscles
* Blood, urine, and skin biopsy samples for testing and sample collection
* After the initial visit, participants will have three more visits, once each in the following 3 years.

DETAILED DESCRIPTION:
Objective

Primary lateral sclerosis (PLS) and amyotrophic lateral sclerosis (ALS) are motor neuron disorders with different phenotypes that progress at very different rates. ALS is a rapidly progressive disease with a median survival less than 5 years. Patients with PLS have a slowly progressive course with a normal lifespan. One hypothesis is that oxidative stress affects the way in which different motor neuron disorders progress. To test this hypothesis, exposures to putative triggers of oxidative stress and biomarkers that may reflect oxidative stress will be assessed in patients with motor neuron disorders. A multicenter effort (the COSMOS study) has been initiated to accumulate sufficient numbers of ALS patients to address this hypothesis. As an add-on study, PLS patients will also be assessed in the multicenter effort. The objective of this protocol is to enroll PLS patients in this multicenter effort. The goal is to assess environmental factors and markers of oxidative stress in patients with established PLS.

Study Population

15 adult patients with PLS who have symptoms of pure upper motor neuron dysfunction for at least 5 but not more than 15 years.

Design

Patients will undergo a standard battery of clinical, physiological, and cognitive screening tests at enrollment, with scheduled follow-up evaluation visits every 12 months for 36 months. Blood and urine samples will be sent to collaborators at Columbia University for analysis of markers of oxidative injury and genetic risk factors. Patients will complete a self-administered nutritional survey and will be interviewed by phone by Columbia University investigators using questionnaires to assess environmental, occupational, lifestyle and psychosocial factors thought to be triggers of oxidative stress.

Outcome Measures

The Columbia University collaborators will combine data from several centers in a regression model correlating the slope of decline of the ALS-FRS score with an index of oxidative stress.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients will be included if they:

Are 20 years or older

Have PLS, that is pure UMN dysfunction (spasticity, pathological hyperreflexia, pathological reflexes with or without motor weakness) of undetermined etiology

Have been evaluated at NIH and are being willing to return for active follow-up for 3 years

Had PLS symptom onset at least 5 years prior to the study enrollment but not more than 15 years

Have normal nerve conduction studies and normal needle electrode examination performed within 12 months of the time of enrollment in this study

Have no other definable diseases causing spasticity such as structural brain or spinal cord disease, metabolic diseases, paraneoplastic syndromes, hereditary diseases, infectious diseases, or other significant neurological abnormalities

Have a reliable family caregiver who can assist in providing responses on telephone interviews and questionnaires if the proband has problems with speaking or writing

Are fluent in English

Ability to provide his/her own informed consent

EXCLUSION CRITERIA:

Patients will be excluded if they:

Have EMG evidence of active denervation or fasciculations in more than a few muscles with chronic neurogenic motor unit potentials at the time of enrollment

Have only lower extremity involvement

Have major medical diseases (e.g. active cancer, dialysis) that have required active medical treatment within the past 6 months

Are participating in clinical treatment trials at the time of enrollment and acquisition of baseline biological samples (participation in clinical trials after the baseline visit is permitted)

Are unwilling or unable to return for follow-up visits

Have pacemakers or other implanted electrical devices, which might make TMS unsafe will be excluded from TMS testing

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-05-13; Study Completion 2015-08-03

PRIMARY OUTCOMES:
Decline in ALSFRS score

CONTACTS AND LOCATIONS:
Overall Officials: Mary Kay Floeter, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gordon PH, Cheng B, Katz IB, Mitsumoto H, Rowland LP. Clinical features that distinguish PLS, upper motor neuron-dominant ALS, and typical ALS. Neurology. 2009 Jun 2;72(22):1948-52. doi: 10.1212/WNL.0b013e3181a8269b. PMID 19487653
- [Background] Strong MJ, Gordon PH. Primary lateral sclerosis, hereditary spastic paraplegia and amyotrophic lateral sclerosis: discrete entities or spectrum? Amyotroph Lateral Scler Other Motor Neuron Disord. 2005 Mar;6(1):8-16. doi: 10.1080/14660820410021267. PMID 16036421
- [Background] Tartaglia MC, Rowe A, Findlater K, Orange JB, Grace G, Strong MJ. Differentiation between primary lateral sclerosis and amyotrophic lateral sclerosis: examination of symptoms and signs at disease onset and during follow-up. Arch Neurol. 2007 Feb;64(2):232-6. doi: 10.1001/archneur.64.2.232. PMID 17296839